CLINICAL TRIAL: NCT03486535
Title: Ultrasound-Guided Infraclavicular Brachial Plexus Block Properties in Diabetic and Non-diabetic Patients: A Prospective Observational Study
Brief Title: Infraclavicular Block Properties in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emine Aysu Salviz, MD, MD, Assoc Prof, EDRA, Istanbul University
Other Study IDs: 2018/203
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus; Nerve Block Duration; Pain, Postoperative
Keywords: Diabetes mellitus; Infraclavicular brachial plexus block; Block duration; Time-to-first pain; Postoperative analgesia
MeSH Terms: conditions — Diabetes Mellitus; Pain, Postoperative | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Diabetic patients: Diabetic patients will receive ultrasound-guided infraclavicular brachial plexus blocks (ICBs) with the mixture of 15 mL lidocaine 2% and 15 mL bupivacaine 0.5%.
  Interventions: Drug: Infraclavicular Brachial Plexus Blocks
- Non-diabetic patients: Nondiabetic patients will receive ultrasound-guided infraclavicular brachial plexus blocks (ICBs) with the mixture of 15 mL lidocaine 2% and 15 mL bupivacaine 0.5%.
  Interventions: Drug: Infraclavicular Brachial Plexus Blocks

INTERVENTIONS:
Drug: Infraclavicular Brachial Plexus Blocks — All patients will receive Infraclavicular Brachial Plexus Blocks with the mixture of lidocaine and bupivacaine. This is an observational study, because all patients will receive the same blocks with the same doses of the local anesthetics. The only difference between groups is including patients with or without Diabetes Mellitus diagnosis. The intervention is the same and these patients cannot be randomized. The aim is investigating the effect of this local anesthetic mixture in Diabetic patients.
  Other Names: Same interventions, drugs and concentrations
  Groups: Diabetic patients
Drug: Infraclavicular Brachial Plexus Blocks — All patients will receive Infraclavicular Brachial Plexus Blocks with the mixture of lidocaine and bupivacaine. This is an observational study, because all patients will receive the same blocks with the same doses of the local anesthetics. The only difference between groups is including patients with or without Diabetes Mellitus diagnosis. The intervention is the same and these patients cannot be randomized. The aim is investigating the effect of this local anesthetic mixture in Nondiabetic patients.
  Other Names: Same interventions, drugs and concentrations
  Groups: Non-diabetic patients

SUMMARY:
Background and objectives: The investigators are performing this study to explore whether the presence of diabetes mellitus (DM) will affect the outcomes of infraclavicular brachial plexus blocks (ICBs) in patients undergoing elbow, forearm and hand surgery.

The primary hypothesis is that the sensory block duration will be delaying in diabetic patients.

Methods: Ethics committee approval has been obtained and after written informed consents, 60 patients are planning to be enrolled to the study. Diabetic patients will be included in Group DM and non-diabetics are included in Group NODM. All patients will receive ultrasound-guided ICBs with the mixture of 15 mL lidocaine 2% and 15 mL bupivacaine 0.5%. Our primary outcome is sensory block duration, and secondary outcomes are sensory and motor block onset times, motor block duration, time-to-first-pain (numeric rating scale (NRS)

≥4), postoperative NRS scores and rescue analgesic consumption (NRS) ≥4) through the postoperative first 2 days. All outcomes will be assessed by blind investigators.

DETAILED DESCRIPTION:
Background and objectives: The impact of diabetes mellitus (DM) on the practice of peripheral nerve blocks need to be investigated on human models, besides animal researches. The investigators have been performing this study to explore whether the presence of DM will affect the outcomes of infraclavicular brachial plexus blocks (ICBs) in patients undergoing elbow, forearm, and hand surgery. The primary hypothesis is that the sensory block duration will be delaying in diabetic patients.

Methods: After obtaining ethics committee approval and written informed consent, 60 patients with American Society of Anesthesiologists (ASA) physical status I-IV and aged between 40 and 80 years are enrolled to the study. Diabetic patients will be included in Group DM and non-diabetics will be included in Group NODM. All patients will receive ultrasound-guided ICBs with the mixture of 15 mL lidocaine 2% and 15 mL bupivacaine 0.5%. Postoperatively, patients will be administered diclomec SR 75 mg IM first and if still needed tramadol 100 mg IV as rescue analgesics (numeric rating scale (NRS) is ≥4). Our primary outcome is sensory block duration, and secondary outcomes are sensory and motor block onset times, motor block duration, time-to-first-pain (numeric rating scale (NRS) ≥4), postoperative NRS scores, and rescue analgesic consumption through the postoperative first 2 days. All outcomes will be assessed by blind investigators.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for arm, elbow, forearm, and hand surgery American Society of Anesthesiologists (ASA) physical status I-IV No regional anesthesia contraindication

Exclusion Criteria:

Type 1 DM, Type 2 DM patients with only 'diet-controlled' therapy Difficulty with understanding the block and follow-up instructions Significant neurologic disorders Psychiatric or cognitive disorders History of substance abuse Acute and/or chronic opioid use Local anaesthetic hypersensitivity or allergy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for arm, elbow, forearm, and hand surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Sensory block duration | 0-24 hours
  Time interval between a successful block (0: full sensation, 1: less sensation, and 2: no sensation) (≥7/8) and the complete restoration of all the senses controlled by the radial, ulnar, median and musculocutaneous nerves (0/8)

SECONDARY OUTCOMES:
Sensory block onset time | 0-30 minutes
  Physical examination with pin-prick test until the block onset (0: full sensation, 1: less sensation, and 2: no sensation) (≥7/8)
Motor block onset time | 0-30 minutes
  Physical examination with modified Bromage scale until the block onset (0: normal motor function; 1: partial motor block, able to flex the elbow and move the fingers but unable to raise the extended arm; 2: almost complete motor block, unable to flex the elbow but able to move the fingers; and 3: complete motor block, unable to move the arm, elbow, or fingers) (≥9/12)
Motor block duration | 0-24 hours
  Time interval between a successful block (0: normal motor function; 1: partial motor block, able to flex the elbow and move the fingers but unable to raise the extended arm; 2: almost complete motor block, unable to flex the elbow but able to move the fingers; and 3: complete motor block, unable to move the arm, elbow, or fingers) (≥9/12) and the complete restoration of all motor responses controlled by the radial, ulnar, median and musculocutaneous nerves (0/12).
Time-to-first pain | 0-48 hours
  Postoperative first pain (Numeric rating scale (NRS) ≥4) (0: no pain, 10: worst pain imaginable)
Pain (NRS) scores | 0-48 hours
  Numeric rating scale (Numeric rating scale (NRS) ≥4) pain scores (0: no pain, 10: worst pain imaginable)
Rescue analgesic consumption | 0-48 hours
  Used postoperatively if (Numeric rating scale (NRS) ≥4) (0: no pain, 10: worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Emine A Salviz, Principal Investigator — Istanbul University, Medical Faculty of Istanbul
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University, Medical Faculty of Istanbul, Istanbul
  - Metin Sabancı Baltalimanı Kemik Hastalıkları Training and Research Hospital, Istanbul

REFERENCES:
- [Result] Salviz EA, Onbasi S, Ozonur A, Orhan-Sungur M, Berkoz O, Tugrul KM. Comparison of Ultrasound-Guided Axillary Brachial Plexus Block Properties in Diabetic and Nondiabetic Patients: A Prospective Observational Study. J Hand Surg Am. 2017 Mar;42(3):190-197. doi: 10.1016/j.jhsa.2017.01.009. PMID 28259276
- [Result] Cuvillon P, Reubrecht V, Zoric L, Lemoine L, Belin M, Ducombs O, Birenbaum A, Riou B, Langeron O. Comparison of subgluteal sciatic nerve block duration in type 2 diabetic and non-diabetic patients. Br J Anaesth. 2013 May;110(5):823-30. doi: 10.1093/bja/aes496. Epub 2013 Jan 24. PMID 23348203